CLINICAL TRIAL: NCT06832280
Title: Improving Parental Support in Hypospadias Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 24-1612; 1R01DK140178-01 (NIH)
Record Dates: First submitted 2025-02-07; First posted 2025-02-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Hypospadias
Keywords: Hypospadias; Pediatric Urologists
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Intervention Model Description: The study team will use block randomization (i.e., four treatment assignments per block) to assign participants to the intervention or control group, stratifying by study site. The full description of the invention vs control arms will be registered after data collection is completed to preserve the scientific integrity of the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Certain members of the research team will also be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Hypospadias Education (Experimental): The parents randomized to this cohort will receive access to an educational website about hypospadias developed by the study team.
  Interventions: Other: Educational Website Developed by Study Team
- Basic Hypospadias Education (Sham Comparator): Parents randomized into the control arm will receive access to a basic educational website about hypospadias.
  Interventions: Other: Basic Educational Website

INTERVENTIONS:
Other: Educational Website Developed by Study Team — This website was developed by the study team in previous research studies.
  Arms: Enhanced Hypospadias Education
Other: Basic Educational Website — This website is a basic education website about hypospadias.
  Arms: Basic Hypospadias Education

SUMMARY:
The proposed study will enroll parent-child pairs and is designed to obtain new knowledge and improve hypospadias care. Parent-child pairs will be randomized into different groups over 36 months and participate for at least 6 months.

DETAILED DESCRIPTION:
The proposed study will approach and enroll parent-child dyads to receive one of two educational websites about hypospadias, a condition that their child has or may have. The parents will be approached and consented before their upcoming consultation with a pediatric urologist regarding hypospadias. The child may have one or more consultation visits with the pediatric urologist. Before the first consultation, the parents will be asked about their current hypospadias knowledge, questions about how they typically interact with doctors, comfort with information presented in a healthcare setting and demographics and then receive access to one of the educational websites. After reviewing the website, the parent will complete a pre-consultation survey asking about hypospadias knowledge and other items. The 1 or 2 urology clinic consultation visits then occur and are optionally audio recorded. After the consultation visit, if the child was found to have no evidence of hypospadias, the child may no longer meet eligibility criteria for the study and may be asked to complete one final telephone call. If the child was otherwise diagnosed with hypospadias, after the final urology consultation visit, the parent will complete the post consultation survey, which consists of questions regarding hypospadias knowledge, care management options, and the treatment chosen. Parents may also be asked to complete an additional phone call regarding any challenges experienced with the website and suggestions for improvement. The final follow up survey will be about 6 months after the treatment decision has been made and will again discuss the treatment option chosen, now that some time has passed.

Pediatric urologists from the two study sites will be asked permission to record their clinic consultations, if the participant family agrees as well.*

*To preserve scientific integrity certain details of the record are not included in the registration, and will be added to the record after the relevant data are gathered.

ELIGIBILITY:
Inclusion Criteria

A parent must meet all of the following criteria to be included:

* Age ≥ 18 years old
* Fluent and literate in English or Spanish
* Parent or legal guardian
* Ability to consent
* One eligible parent per child
* Plan to attend urology consultation
* Has access to a smart phone, tablet, or computer with reliable internet access
* Has the ability and agrees to receive unencrypted communications by text or email

A child must meet all of the following criteria to be included:

* 0-5 years old at the time of urology consultation
* Have an upcoming urology consult with an enrolled pediatric urologist regarding hypospadias

Exclusion Criteria

If a parent meets any of the following criteria they will be excluded:

* Previous participant in hypospadias study
* Parent has another child with hypospadias or father of the child has a known history of hypospadias
* Parent is unaware of any penile abnormality with child
* A final hypospadias treatment decision has been made in discussion with a pediatric urologist
* Investigator discretion

If a child meets any of the following criteria they will be excluded:

* Prior hypospadias surgery
* Upcoming hypospadias urology consult scheduled less than a week away from when the patient was identified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-07-25 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean primary outcome measure 1 score (to be disclosed after final subject completes T3 data collection)* | Post-clinic visit, 1-30 days after the final clinic visit (T3)
  Measures primary outcome 1 construct.
  The total possible range of scores is from 1 to 6, where higher scores indicate more of the primary outcome 1 construct.
  *To preserve scientific integrity certain details of the record are not included in the registration and will be added to the record after all primary outcome data have been gathered.
Mean primary outcome measure 2 score among 50% of participants (to be disclosed after final subject completes T3 data collection)** | Clinic visit(s), 3-60 days after enrollment (T2a) and up to 12 months after the first clinic visit (T2b). Note some patients will only have T2a.
  Clinic visits will be audio recorded and coded using primary outcome measure 2 to measure primary outcome 2 construct.
  The total possible range of scores is from 0 to 4, where higher scores indicate more of the primary outcome 2 construct.
  **To preserve scientific integrity certain details of the record are not included in the registration and will be added to the record after all primary outcome data have been gathered.

SECONDARY OUTCOMES:
Mean visit duration among 50% of participants | Clinic visit(s), 3-60 days after enrollment (T2a) and up to 12 months after the first clinic visit (T2b). Note some patients will only have T2a.
  Time stamps from audio recorded clinic visits will be used to calculate visit duration in minutes.
  The total possible range of duration is estimated to be 10 to 40 minutes. Higher numbers indicate longer duration.
Mean change in Low Literacy Decisional Conflict Scale (DCS-LL) scores (T1-T0, T3-T0, and T3-T1) | Baseline, 3-60 days before the first clinic visit (T0) Pre-clinic visit, 1-7 days before the first clinic visit (T1) Post-clinic visit, 1-30 days after the final clinic visit (T3)
  The DCS-LL measures the degree of decisional conflict.
  The total possible range of scores is from 0 to 100 with higher scores indicating more conflict.
Mean change in Hypospadias Knowledge Assessment scores (T1-T0, T3-T0, and T3-T1) | Baseline, 3-60 days before the first clinic visit (T0) Pre-clinic visit, 1-7 days before the first clinic visit (T1) Post-clinic visit, 1-30 days after the final clinic visit (T3)
  Measures hypospadias knowledge.
  The total possible range of scores is from 0 to 6 with higher scores indicating more knowledge.
Mean score on Decisional Regret Scale | Follow-up (T4): 150-210 days post-final clinic visit in non-surgery patients;150-210 days postoperatively in surgery patients. Because surgery may occur up to 18 months after the last clinic visit, not all participants will complete T4 before study end
  Measures distress/remorse after a healthcare decision.
  The total possible range of scores is from 1 to 5 with higher scores indicating more regret.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Schilling, MD, MSHP, Principal Investigator — UNC Chapel Hill
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data collected during the trial will be deposited in the UNC Dataverse, a trustworthy, generalist data repository managed by the Research Data Management Core at the University of North Carolina at Chapel Hill. UNC Dataverse provides persistent identifiers, robust standardized metadata, and is committed to long-term preservation and access of research data. Data are published under a CC0 license by default with customizable terms of use as needed. Additionally, UNC Dataverse is routinely backed up and preserved on multiple geographically distributed servers and is a member of Data-PASS, a community committed to the sustainability and access of research data.
Supporting Information: Study Protocol
Time Frame: Beginning 36 months (3 years) following article (primary aim) publication and ending 60 months (5 years) following article publication.
Access Criteria: Data will be shared with researchers who (1) provide a methodologically sound proposal that focuses on meta-analysis, (2) have obtained IRB approval for the proposal, and (3) execute a data use agreement.
  Proposals should be directed to Samantha_Schilling@med.unc.edu and improvinghypocare@unc.edu.
URL: https://researchdata.unc.edu/dataverse-information/